CLINICAL TRIAL: NCT02868580
Title: Phase 2a Open Label Study, Safety and Tolerability of Combination Antiretroviral Therapy (Triumeq) in Participants With Amyotrophic Lateral Sclerosis (ALS) - The Lighthouse Project.
Brief Title: Safety and Tolerability of Antiretroviral (Triumeq) in Patients With Amyotrophic Lateral Sclerosis (ALS).
Acronym: Lighthouse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuroscience Trials Australia (Other)
Collaborators: Macquarie University, Australia (Other); Westmead Hosptial (Unknown); Calvary Health Care Bethlehem (Unknown); The University of Sydney - Brain and Mind Centre (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUR-101
Record Dates: First submitted 2016-06-16; First posted 2016-08-16 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Antiretroviral Therapy, Triumeq
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — abacavir, dolutegravir, and lamivudine drug combination; dolutegravir; abacavir; Lamivudine

STUDY DESIGN:
Intervention Model Description: Safety and Tolerability open label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm open label (Experimental): All subjects will receive open label Triumeq following a lead-in phase. Triumeq is abacavir 600mg, lamivudine 300mg, dolutegravir 50mg
  Interventions: Drug: Triumeq

INTERVENTIONS:
Drug: Triumeq — Triumeq, a combination of dolutegravir, abacavir and lamivudine is an anti-retroviral therapy indicated for people with HIV-1 infection.
  Other Names: dolutegravir (50mg); abacavir (600mg); lamivudine (300mg)

SUMMARY:
This is a phase 2a open label, multicentre design study to investigate the safety of Triumeq in patients with ALS at 24 weeks post treatment. In this phase 2a study the investigators aim to determine whether a combination of anti-retroviral therapy, Triumeq (dolutegravir 50mg, abacavir 600mg, lamivudine 300mg) is tolerated and safe in patients with ALS. As secondary outcomes, ALSFRS-R, ALSQOL, physical examination, neurophysical parameters and respiratory and muscle function will be evaluated. Blood and urine samples will be stored for possible future analysis for viral activity. Subjects will be screened for the study after signing an approved Informed consent document.

DETAILED DESCRIPTION:
This study will be a multi-centre, open-label longitudinal study to investigate the safety and tolerability of combination antiretroviral therapy (Triumeq) in Motor Neuron Disease (MND)/Amyotrophic Lateral Sclerosis (ALS) for 24 weeks in 40 HIV negative ALS patients.

The overall study duration will be 34 weeks, with up to 14 days for screening, followed by an 8-week lead-in phase and 24-week treatment phase. Outcomes will be measured at 4, 8, 12, 20 and 24 weeks. Participants will be followed at 4-weekly intervals for safety and clinical measures.

Subjects will be screened for the study after signing an approved Informed consent form. As part of the 14 day screening phase, subjects will undertake an extensive medical and neurological assessments.

Following the screening phase subjects will enter the 8 week lead-in-phase. During this phase, they will undertake two ALSFRS-R at 4 week intervals. The ALSFRS-R will be undertaken with the subject by telephone.

At the baseline visit, following the lead-in-period, blood and urine will be taken for safety monitoring and also bio-banked for possible future measurement of Human Endogenous Retroviruses (HERVs). Baseline signs and symptoms will be collected.

All subjects will have their inclusion and exclusion criteria checked at the Baseline visit (Week 0) and eligible subjects will start the Triumeq.

Subjects will return to the centre on Weeks 4, 8, 16, 24 and at 7 days after the last dose of investigational product (or early termination) to undertake a neurological examination as well as an assessment of the ALS Functional Rating Scale-Revised (ALSFRS-R), neurophysical index (NPI), forced vital capacity (FVC) as measured by handheld spirometer, SNIP test and quantitative hand muscle testing by dynamometry. All subjects will undertake an evaluation of hematological and biochemical parameters and collection of blood and urine samples for bio-banking. A voice recording will be undertaken.

At early termination visit, subjects will undergo an ECG Test. At baseline, weeks 8, 16 and 24 or early termination visit subjects will be asked to complete the Columbia Suicide Severity Rating Scale. At screening week 8 and end of treatment/early termination visit, subjects will also be asked to complete an ALSFRS-R.

SAE's, AE's and changes to concomitant medications will be observed and evaluated throughout the study. Each study visit will have a 7 day window after the due date to account for scheduling conflicts/holidays/weekends.

Subjects will be given additional study product to account for the 7- day window.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be eligible to participate in this study:

* Age 18-75 years at the time of the screening visit
* Able to provide informed consent and comply with study procedures
* Sporadic ALS diagnosed as probable, laboratory-supported probable or definite according to the World Federation of Neurology El Escorial revised criteria as determined by a neurologist with neuromuscular sub-specialty training
* Diagnosis <24 months from date of enrolment
* (Forced) Vital capacity at least 60% of predicted value for gender, height and age at the screening visit
* Must be on a stable dose of riluzole for at least 30 days prior to the screening visit.
* Subject has established care with a neurologist at one of the four specialized ALS clinics involved in the study and will maintain this clinical care throughout the study.
* Subjects can participate in clinical registries, but will be excluded to this protocol if they are participating in a clinical trial involving additional or investigative treatment exposure.

Exclusion Criteria:

A participant will be excluded if he or she has any of the following:

* Dependence on mechanical ventilation at the time of screening
* Gastrostomy at the time of screening
* Absence of Upper Motor Neuron Signs
* Participation in any other investigational drug trial or using investigational drug (within 12 weeks prior to screening)
* Known hypersensitivity to dolutegravir, abacavir or lamivudine, or to any of the excipients
* Presence of the HLA-B*5701 allele at screening
* Presence of a monogenic cause of ALS (e.g. known mutation in SOD1, expansion in c9orf72 etc.)
* History of positive test or positive result at screening for HIV
* Subjects positive for Hepatitis B at screening (+HBsAg), or anticipated need for Hepatitis C virus (HCV) therapy during the study*;
* Women must not be able to become pregnant (post menopausal for >1 year, surgically sterile, adequate contraception) or breastfeed for the duration of the study. Women of childbearing potential must have a negative pregnancy test at screening and be non-lactating
* Other interventional clinical trial
* Subject is taking medication contraindicated with Triumeq. Dofetilide (or pilsicainide [available in Japan]) is prohibited as DTG may inhibit its renal tubular secretion resulting in increased dofetilide concentrations and potential for toxicity.
* Presence of any of the following clinical conditions at the time of screening:

Drug or alcohol abuse Unstable medical disease (such as unstable angina or chronic obstructive pulmonary disease), or active infectious disease (such as Hepatitis B or C or tuberculosis), or current malignancy Unstable psychiatric illness defined as psychosis or untreated major depression within 90 days of the screening visit. This exclusion criteria is based on a prior psychiatric diagnosis that is unstable as determined by the subject's treating Psychiatrist Dementia as previously diagnosed by a medical practitioner

• Safety Laboratory Criteria at the screening visit: Alanine aminotransferase (ALT) >5 times the upper limit of normal (ULN), OR ALT >3xULN Total bilirubin, lactate, triglycerides, amylase, or lipase greater than 2.0 times the upper limit of normal Subject has creatinine clearance of <50 mL/min via Cockroft-Gault method Subjects with moderate to severe hepatic impairment (Class B or greater) as determined by Child-Pugh classification; Absolute neutrophil count of < 1 x 109/L Platelet concentration of < 100 x 109/L Haemoglobin < 100g/L

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment related adverse events as defined CTCAE V4.0. | 1 year
  Safety will be measured by Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment.

SECONDARY OUTCOMES:
ALS Functional Rating Scale-Revised (ALSFRS-R) scoring | 1 year
  Efficacy will be measured by the change in scores of the ALS Functional Rating Scale-Revised (ALSFRS-R) conducted at screening, twice within the lead-in phase and at four weekly intervals during the study until end of treatment or early termination.
Number of Participants With Abnormal Laboratory Values for Neurophysiological Index (NI) Related to Treatment. | 1 year
  A neurophysiological index (NI) measurement will be calculated according to the parameters of Compound Muscle Action Potential amplitude/DML x Frequency % to determine the index score.
Number of participants with abnormal Sniff Nasal Inspiratory Pressure (SNIP) Test results | one year
  The SNIP test results will be calculated according to the Pn(sn) as a percentage of predicted value according to treatment.
Number of participants with abnormal forced vital capacity (FVC) test results as measured by hand-held spirometry | One year
  The FVC test results will be measured in liters and reported according to percentage of predicted values for participants on treatment
Number of participants with abnormal quantitative hand muscle testing as measured by dynanometry. | One year
  The quantitative hand muscle strength will be assessed by 3 Measurements on Grip Strength and Pinch Grip: measurement in kilograms
Number of participants with abnormal scores on the Columbia Suicide Severity Score C-SSRS). | One year
  The C-SSRS is a measure of suicidal ideation and behavior. It is a composite numerical scale divided into sections and used to assess selected parameters over time in participants on treatment. The scoring system is both binomial and rating scale and is reported according to different aspects of the assessment.

OTHER OUTCOMES:
Number of participants with abnormal ECG results | one year
  ECGs will be performed at screening, 16 and 24 weeks and early termination for participants on treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Gold, MD, Principal Investigator — The Albion Centre
Locations (4):
- Australia (4):
  - Macquarie Neurology, North Ryde, New South Wales
  - Westmead Hospital, Parramatta, New South Wales
  - Brain and Mind Centre, Sydney, New South Wales
  - Calvary Health Care Bethlehem, Caulfield South, Victoria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ramirez P, Zuniga G, Sun W, Beckmann A, Ochoa E, DeVos SL, Hyman B, Chiu G, Roy ER, Cao W, Orr M, Buggia-Prevot V, Ray WJ, Frost B. Pathogenic tau accelerates aging-associated activation of transposable elements in the mouse central nervous system. Prog Neurobiol. 2022 Jan;208:102181. doi: 10.1016/j.pneurobio.2021.102181. Epub 2021 Oct 17. PMID 34670118